CLINICAL TRIAL: NCT00043992
Title: Outdoor Allergen Exposure, Sensitivity, and Acute Asthma
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Other Study IDs: 9744-CP-001
Record Dates: First submitted 2002-08-16; First posted 2002-08-19 (Estimated); Last update posted 2006-09-04 (Estimated); Status verified 2006-09

CONDITIONS: Asthma
Keywords: Asthma; Allergens
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
To examine the role of outdoor pollen grains and fungal spores in the exacerbation of asthma and to produce forecasting models to predict days of high concentration.

DETAILED DESCRIPTION:
Asthma is a growing problem, and outdoor allergens play a role in exacerbation of many cases. A clearer understanding of this role and its magnitude, and a means of controlling the effects of outdoor allergen exposures is needed. We propose Poisson time-series and conditional panel studies to test these hypotheses: 1) The incidence of acute asthma attacks, as measured by urgent care inhalation treatments and hospitalizations for asthma, has a dose-dependent relationship with exposure to specific outdoor allergens; 2) Specific sensitization to outdoor allergens is a risk factor for having an acute attack; and 3) Exposure conditions that lead to acute asthma attacks can be forecast, creating an opportunity to reduce asthma morbidity and mortality ny targeting pretreatment and/or exposure controls.

ELIGIBILITY:
Must be a member of the Fallon HMO and be treated for acute asthma exacerbation.

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1000
Dates: Start 2001-07

CONTACTS AND LOCATIONS:
Locations (1):
- Fallon Clinic and Fallon Community Health Plan, Worcester, Massachusetts, United States